CLINICAL TRIAL: NCT01155258
Title: Phase I Clinical Trial of Temsirolimus and Vinorelbine in Advanced Solid Tumors.
Brief Title: Temsirolimus and Vinorelbine Ditartrate in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-09-6; NCI-2010-01382
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Hereditary Paraganglioma; Male Breast Cancer; Malignant Paraganglioma; Metastatic Gastrointestinal Carcinoid Tumor; Metastatic Pheochromocytoma; Pancreatic Polypeptide Tumor; Recurrent Breast Cancer; Recurrent Cervical Cancer; Recurrent Endometrial Carcinoma; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Recurrent Neuroendocrine Carcinoma of the Skin; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pheochromocytoma; Recurrent Prostate Cancer; Recurrent Renal Cell Cancer; Recurrent Small Cell Lung Cancer; Recurrent Uterine Sarcoma; Regional Gastrointestinal Carcinoid Tumor; Regional Pheochromocytoma; Stage III Cervical Cancer; Stage III Endometrial Carcinoma; Stage III Neuroendocrine Carcinoma of the Skin; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage III Prostate Cancer; Stage III Renal Cell Cancer; Stage III Uterine Sarcoma; Stage IIIA Breast Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Breast Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Endometrial Carcinoma; Stage IV Neuroendocrine Carcinoma of the Skin; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Prostate Cancer; Stage IV Renal Cell Cancer; Stage IV Uterine Sarcoma; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Paraganglioma, Extra-Adrenal; Pheochromocytoma; Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Islet Cell; Carcinoma, Merkel Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Prostatic Neoplasms; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Carcinoma, Medullary | interventions — temsirolimus; Sirolimus; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and vinorelbine ditartrate IV over 5-10 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Drug: vinorelbine ditartrate

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; rapamycin analog CCI-779; Torisel
Drug: vinorelbine ditartrate — Given IV
  Other Names: Biovelbin; Eunades; navelbine ditartrate; NVB; vinorelbine tartrate; VNB

SUMMARY:
RATIONALE: Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vinorelbine ditartrate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus together with vinorelbine ditartrate may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of giving temsirolimus and vinorelbine ditartrate together in treating patients with unresectable or metastatic solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerated dose (MTD) for the combination of temsirolimus and vinorelbine in advanced solid tumors.

II. To obtain preliminary information regarding the activity of this combination.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of this combination.

OUTLINE:

Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and vinorelbine ditartrate IV over 5-10 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion

* Patients with histologically confirmed metastatic or unresectable solid tumors for which standard curative measures do not exist or are no longer effective; histology will be limited to those tumors for which temsirolimus or vinorelbine have reported clinical activity: lung, breast, ovary, cervix, prostate, uterus, renal, bladder and neuroendocrine tumors
* SWOG performance status of 0-2
* Projected life expectancy of at least 3 months
* Provision of informed consent prior to any study-related procedures
* Negative pregnancy test for women of childbearing potential
* Female patients must not be pregnant due to the potential mutagenicity and teratogenicity of this treatment; a pregnancy test must be administered 7 days prior to administration of therapy to women of childbearing potential; patients must agree to use some form of contraception while on this study at initiation and for the duration of participation in the study; sexually active males must also use a reliable and appropriate method of contraception; post-menopausal women must be amenorrheic for at least 12 months to be considered of nonchildbearing potential
* Patients must have recovered from acute toxicities from previous surgery, chemotherapy or radiation therapy
* ANC >= 1500/mm^3
* Platelet count >= 100,000 cells/mm^3
* Hemoglobin >= 9.0g/dL
* Serum creatinine =< 1.5 mg/dl
* Hepatic function: Patients must have adequate liver functions: AST or ALT =< 2.5 X upper limit of normal (ULN), alkaline phosphatase =< 2.5 X upper limit of normal; in patients with bone metastasis and no evidence of liver metastasis and bilirubin =< upper limit of normal an alkaline phosphatase =< 5 ULN will be allowed
* Serum Bilirubin =< 1.0 mg/dL
* Peripheral neuropathy grade 0-1
* No other concomitant therapy directed at the cancer is allowed

Exclusion

* Prior therapy with vinorelbine or an mTor inhibitor
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Last dose of prior chemotherapy discontinued less than 4 weeks before the start of study therapy
* Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy
* Any unresolved toxicity greater than CTC grade 1 from previous anticancer therapy, excluding alopecia
* CTC Grade 1 or greater neuropathy (motor or sensory) at study entry
* Hematologic function with absolute neutrophils =< 1500/mm^3 and/or platelets < 100,000/mm^3
* Hepatic function with serum bilirubin greater than the upper institutional limits of normal, ALT and AST > 2.5 times the upper institutional limits of normal
* Concurrent use of strong inhibitors of CYP3A4: ketoconazole, itraconazole, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine and voriconazole
* CYP3A4 inducers should be avoided or used with caution; the use of these agents is discouraged: rifabutin, rifampicin, rifapentine, carbamazepine, Phenobarbital, phenytoin and St. John's wart
* Ongoing long term use of steroids for chronic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of Temsirolimus and Vinorelbine | 1 month up to 18 months
To assess the response rate based on the Response Evaluation Criteria in Solid Tumors (RECIST) | 2 months up to 18 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Temsirolimus and Vinorelbine | 4 weeks up to 36 weeks
Progression-free and overall survival | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States